CLINICAL TRIAL: NCT04189965
Title: Traumatic Long-term Memory of Pain - Pain Conditioning Study in Humans
Brief Title: Traumatic Long-term Memory of Pain in Humans
Acronym: TRAUMADOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL19_0413
Record Dates: First submitted 2019-11-22; First posted 2019-12-09 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Pain; Traumatic Memory
Keywords: Pain; Traumatic Long-term Memory
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilot group (Other): Subjects are volunteers of 18 to 50 years of age that have given consent and that are affiliated to a social security. Overall, subjects must be in good health (no chronic pain, neuropathy or cardiac/respiratory issues etc.) and (for women) non-pregnant.
  The subject will be seated in an armchair. He will be asked to explore the virtual environment using virtual reality glasses to validate it.
  The subject will also have headphones and different shouts or noises will be broadcast and he will have to rate the level of dislike of each sound stimulation.
  Interventions: Other: Validation of virtual environment and auditive stimulation with virtual reality glasses (Pilot phase)
- Experimental group (Other): Subjects are volunteers of 18 to 50 years of age that have given consent and that are affiliated to a social security. Overall, subjects must be in good health (no chronic pain, neuropathy or cardiac/respiratory issues etc.) and (for women) non-pregnant.
  The subject will be seated in an armchair. He will be asked to explore the virtual environment using virtual reality glasses. He will also have headphones and different shouts or noises will be broadcast and an electric stimulation glove to study in humans the mechanisms of long-term memory of pain by exploring the parallel between memory of pain and memory of a traumatic event.
  3 sessions of stimulation will be done (D0, D2 and D30)
  Interventions: Other: Electrical cutaneous stimulation and auditive stimulation (Principal Experimental phase)
- Experimental subgroup (Other): Subjects are volunteers of 18 to 50 years of age that have given consent and that are affiliated to a social security. Overall, subjects must be in good health (no chronic pain, neuropathy or cardiac/respiratory issues etc.) and (for women) non-pregnant.
  The subject will be seated in an armchair. He will be asked to explore the virtual environment using virtual reality glasses. He will also have headphones and different shouts or noises will be broadcast and an electric stimulation glove to study in humans the mechanisms of long-term memory of pain by exploring the parallel between memory of pain and memory of a traumatic event.
  3 sessions of stimulation will be done (D0, D2 and D30)
  Interventions: Other: Electrical cutaneous stimulation and auditive stimulation (Secondary Experimental phase)

INTERVENTIONS:
Other: Validation of virtual environment and auditive stimulation with virtual reality glasses (Pilot phase) — The goal of this phase is the development of the experimental protocol in virtual reality. Virtual environment will be checked and auditive stimulation will be graduated.
  Arms: Pilot group
Other: Electrical cutaneous stimulation and auditive stimulation (Principal Experimental phase) — This phase is the principal step of the study: during moving in virtual environment, electrical stimulation on one hand and auditive stimulation will be applied. EEG, ECG and skin conductance will be measured during conditioning phase and extinction phase (day 1, 30 minutes each phase). Behavioral measures will be done throughout the 3 sessions (day 1, day 2 and day 30)
  Arms: Experimental group
Other: Electrical cutaneous stimulation and auditive stimulation (Secondary Experimental phase) — This phase is the same of the Principal Experimental phase except for the EEG that will not be performed.
  Arms: Experimental subgroup

SUMMARY:
Few studies have focused on understanding the mechanisms underlying pain memory in humans. Thus, this project aims to investigate the link between pain memorisation and memorisation of the associated context by addressing the issue of pain conditioning. The study is composed of two successive parts: one pilot then one experimental. The goal is to understand pain memorisation processes by analysing the parallel between pain memorisation and memorisation of a traumatic event. By using immersive virtual reality, investigators aim to show that contextual pain conditioning is associated with : 1- a specific neural networks; 2- a reactivation of vegetative and behavioural reactions related to pain as well as electro-physiological markers when re-exposure to the specific pain-conditioning-context; 3- an implicit hypermnesia of the pain-associated context and a struggle to extinguish conditioning; 4- a favoured elaboration of false memories of the contextual pain. The emitted hypothesis suggests that a cortical and behavioural mnemonic trace is created during encoding of pain in association with its context, and that the latter can reactivate although the pain itself has disappeared. This implicit cortical mnemonic trace, evoked by the simple pain-associated context, could explain the notion of pain print persisting at long-term in patients suffering from chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Subject between 18 and 50 years old
* Subjects having given their written consent
* Subjects with health insurance

Exclusion Criteria:

* Prior addiction to drugs
* Prior neurological issues
* Chronic pain (neuropathic or non-neuropathic)
* Pregnant/breast-feeding women
* Absence of efficient contraception method for the duration of the study (1 month) for participants of procreation age (no inclusion limitation for male participants of procreation age)
* Subjects under chronic analgesic treatment or having taken an analgesic treatment in the 24 h preceding the experiment
* Heart issues
* Subjects under justice surveillance
* Subjects participating in another study which inclusion period overlaps with the one from this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Measurement of electrophysiological (EEG) changes during a pain conditioning set up and its extinction | day 1
  The EEG will be done throughout the conditioning phase and the extinction phase (30 minutes each)conducted during the first session of the experiment (Day 1)
Measurement of vegetative (electrodermal, electrocardiac) changes during a pain conditioning set up and its extinction | day 1
  The cutaneous response and electro-cardiographic activity will be done throughout the conditioning phase and the extinction phase (30 minutes each)conducted during the first session of the experiment (Day 1)

SECONDARY OUTCOMES:
Assessment of short-term memory of an environment according to whether it is associated with a painful stimulation or not | day 2
  This outcome is evaluated by combined tests:
  * Free recall test: the subjects will have to quote a maximum of memorized objects during the conditioning phase
  * Recognition test: the objects present in the environment as well as objects not present in the environment will be presented randomly on a screen. Subjects should indicate whether the object in question was present in the environment or not.
Assessment of long-term memory of an environment according to whether it is associated with a painful stimulation or not | day 30
  This outcome is evaluated by combined tests:
  * Free recall test: the subjects will have to quote a maximum of memorized objects during the conditioning phase
  * Recognition test: the objects present in the environment as well as objects not present in the environment will be presented randomly on a screen. Subjects should indicate whether the object in question was present in the environment or not.
Assessment subject capacity to create false memory of environment according to the associated stimulation (pain or no pain) | day 2
  Questionnaire will be conducted on environment (presence or absence of different objects) to assess false memories
Assessment subject capacity to create false memory of environment according to the associated stimulation (pain or no pain) | day 30
  Questionnaire will be conducted on environment (presence or absence of different objects) to assess false memories
Eye-tracking measurements, to assess the exploration of different contexts according to their nature | Day 1
  An Eye-tracking system will be included in the Virtual Reality glasses (used during conditioning and extinction) to assess eye-movement during exploration of the environment
Assessment of the total duration needed for total extinction | 30 minutes
  The amount of time needed for vegetative reactions to go back to baseline will be assessed during the extinction phase

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Neurologique,, Bron, France